CLINICAL TRIAL: NCT02202512
Title: Effect of Repeated Oral Doses of BI 1060469, BI 1021958 and Active Controls, Cimetidine and Naproxen, on Measured GFR Via Renal Clearance of Iohexol in Healthy Male Subjects (a Phase I Study; Single-blind, Randomized, Placebo-controlled Within BI Groups and Open-label for the Active Controls)
Brief Title: Effect of Repeated Doses of BI 1060469 and BI 1021958 on Glomerular Filtration Rate (GFR) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1333.43; 2014-000320-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-07-28; First posted 2014-07-29 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Cimetidine; Naproxen

ARMS (5):
- BI 1060469 low dose (Experimental): Low-Dose,Tablet,oral administration with 240 ml water,over 10 days
  Interventions: Drug: Placebo; Drug: BI 1060469 low dose
- BI 1060469 high dose (Experimental): High-Dose,Tablets,oral administration with 240 ml water, over 10 days
  Interventions: Drug: Placebo; Drug: BI 1060469 high dose
- Cimetidine (Active Comparator)
  Interventions: Drug: Cimetidine
- Naproxen (Active Comparator)
  Interventions: Drug: Naproxen
- BI 1021958 (Experimental): High-Dose,Tablets,oral administration with 240 ml water, over 10 days
  Interventions: Drug: Placebo; Drug: BI 1021958

INTERVENTIONS:
Drug: Placebo — tablets
  Arms: BI 1060469 low dose
Drug: Cimetidine
  Arms: Cimetidine
Drug: Placebo — tablets
  Arms: BI 1060469 high dose
Drug: Placebo — tablets
  Arms: BI 1021958
Drug: BI 1060469 high dose — tablets
  Arms: BI 1060469 high dose
Drug: BI 1060469 low dose — tablets
  Arms: BI 1060469 low dose
Drug: Naproxen
  Arms: Naproxen
Drug: BI 1021958 — tablets
  Arms: BI 1021958

SUMMARY:
Main objective is to investigate the measured glomerular filtration rate (mGFR) as assessed by iohexol clearance in healthy male normovolemic subjects after oral administration of single and repeated doses of BI 1060469, and BI 1021958.

The secondary objective of this trial is to investigate the glomerular filtration rate (GFR) as assessed by 24 hours creatinine clearance in healthy male normovolemic subjects after oral administration of single and repeated doses of BI 1060469, and BI 1021958.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigators assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests, including negative test result on occult blood in stool (only for subjects assigned to Naproxen)
* Age 18 to 45 years (incl.)
* Body Mass Index (BMI) 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged clinically relevant by the investigator
* Repeated measurement of systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, or pulse rate outside the range of 50 to 90 mmHg
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Serum creatinine laboratory value out of the normal range
* GFR (Glomerular Filtration Rate) < 90 mL/ min at screening
* Urinary toral protein/creatinine ratio > 0,1 mg protein/ mg creatinine
* Current or history of relevant kidney, urinary tract diseases or abnormalities (i.e. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure, infections)
* Further exclusion criteria may apply

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
measured glomerular filtration rate (mGFR) based on renal iohexol clearance | up to day 11

SECONDARY OUTCOMES:
measured urinary 24-hour creatinine clearance | up to day 11

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1333.43.1 Boehringer Ingelheim Investigational Site, Berlin, Germany